CLINICAL TRIAL: NCT04186429
Title: Epigegenetic Influences on Neurobehavioral Recovery Following Pediatric Traumatic Brain Injury
Brief Title: Epigenetic Effects on Traumatic Brain Injury Recovery
Acronym: EETR
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Amery Treble, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY19040402; 1K01HD097030-01A1 (NIH)
Record Dates: First submitted 2019-11-26; First posted 2019-12-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Traumatic Brain Injury; Orthopedic Injury
Keywords: traumatic brain injury; rehabilitation; neuropsychology; precision medicine; epigenetic; proteomic; brain-derived neurotrophic factor; recovery; neurobehavioral outcomes; children; childhood adversity; biomarkers
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, saliva, cerebrospinal fluid

GROUPS / COHORTS (2):
- traumatic brain injury: Children with traumatic brain injury
- orthopedic injury: Children with orthopedic injury

SUMMARY:
Methylation of the brain-derived neurotrophic factor (BDNF) gene is involved in both the biological encoding of childhood adversity and neuroplasticity following traumatic brain injury (TBI). This research will characterize BDNF methylation during recovery from TBI in children and investigate this novel biomarker as a potential biological mechanism underlying the known association between childhood adversity and poorer neurobehavioral outcomes following TBI in childhood. Findings from this research will contribute to an improved understanding of why some children display good recovery following TBI, whereas many others suffer from chronic neurobehavioral impairments.

DETAILED DESCRIPTION:
Unexplained heterogeneity in outcomes following pediatric traumatic brain injury (TBI) is one of the most critical barriers to the development of effective prognostic tools and therapeutics. The addition of personal biological factors to our prediction models may account for a significant portion of unexplained variance and advance the field towards precision rehabilitation medicine. The overarching goal of the Epigenetic Effects on Pediatric Traumatic Brain Injury Recovery (EETR) study is to investigate an epigenetic biomarker involved in both childhood adversity and post-injury neuroplasticity to better understand heterogeneity in neurobehavioral outcomes following pediatric TBI. The primary hypothesis is that childhood adversity will be associated with poorer neurobehavioral recovery in part through an epigenetically mediated reduction in brain-derived neurotrophic factor (BDNF) expression in response to TBI.

EETR is an observational, prospective, longitudinal concurrent cohort study of children aged 3-18 years with either TBI (n=200) or orthopedic injury (n=100), recruited from the UPMC Children's Hospital of Pittsburgh. Participants complete study visits acutely and at 6- and 12-months post-injury. Blood and saliva biosamples are collected at all time points-and CSF when available acutely-for epigenetic and proteomic analysis of BDNF. Additional measures assess injury characteristics, pre- and post-injury child neurobehavioral functioning, childhood adversity, and potential covariates/confounders. Analyses will characterize BDNF DNA methylation and protein levels over the recovery period and investigate this novel biomarker as a potential biological mechanism underlying the known association between childhood adversity and poorer neurobehavioral outcomes following pediatric TBI.

ELIGIBILITY:
Inclusion criteria:

-hospitalized overnight for a non-penetrating complicated mild to severe TBI as defined by the lowest post-resuscitation Glasgow Coma Scale (GCS) score or orthopedic injury.

Complicated mild TBI is defined as a GCS of 13-15 with neuroimaging indicating intracranial or parenchymal injury or depressed/displaced skull fracture. Moderate TBI is defined as GCS 9-12. Severe TBI is defined as GCS 3-8. Children are included in the OI group if they sustain a bone fracture, excluding to the skull or face, without any signs of head trauma or brain injury (e.g. nausea/vomiting, headache, loss of consciousness, GCS below 15 at any point).

Exclusion criteria:

* non-English-speaking child or non-English-speaking parents/guardians
* documented or parent-reported history of previous TBI/concussion requiring overnight hospitalization
* pre-injury neurological disorder or intellectual disability
* pre-injury psychiatric disorder requiring hospitalization
* sensory or motor impairment precluding study measure completion
* pregnancy at the time of study participation
* participants are also excluded if at least one biosample is not able to be collected within 7 days of the injury

Ages: 3 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children hospitalized overnight at UPMC Children's Hospital of Pittsburgh for complicated mild to severe traumatic brain injury or orthopedic injury.
Sampling Method: Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
NIH Toolbox Cognition Battery (NIHTB-CB) | 6 months post-injury
  The NIHTB-CB is a 30-minute battery of standardized neuropsychological tests administered on an iPad. The NIHTB-CB provides norm-referenced scores for the domains of language, episodic memory, processing speed, working memory, and executive function, as well as an overall cognitive function composite score. Higher T scores indicate better neuropsychological performance.
NIH Toolbox Cognition Battery (NIHTB-CB) | 12 months post-injury
  The NIHTB-CB is a 30-minute battery of standardized neuropsychological tests administered on an iPad. The NIHTB-CB provides norm-referenced scores for the domains of language, episodic memory, processing speed, working memory, and executive function, as well as an overall cognitive function composite score. Higher T scores indicate better neuropsychological performance.
Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) or Preschool Version (BRIEF-P) | 6 months post-injury
  To assess everyday executive functioning, parents complete the Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) or Preschool Version (BRIEF-P). Three composite scores are computed for behavioral regulation, emotion regulation, and cognitive regulation, as well as a global executive composite. Higher T scores indicate poorer executive function.
Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) or Preschool Version (BRIEF-P) | 12 months post-injury
  To assess everyday executive functioning, parents complete the Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) or Preschool Version (BRIEF-P). Three composite scores are computed for behavioral regulation, emotion regulation, and cognitive regulation, as well as a global executive composite. Higher T scores indicate poorer executive function.
Strengths and Difficulties Questionnaire | 6 months post-injury
  The Strengths and Difficulties Questionnaire (SDQ) measures psychological adjustment. Subscales include Emotional Symptoms, Conduct Problems, Hyperactivity-Inattention, Peer Problems, and Prosocial Behavior. A Total Difficulties score is also provided. Four different versions are administered based on the child's age. Higher raw scores on all scales except for Prosocial Behavior indicate more difficulties; higher raw scores on Prosocial Behavior indicate greater prosocial behavior.
Strengths and Difficulties Questionnaire | 12 months post-injury
  The Strengths and Difficulties Questionnaire (SDQ) measures psychological adjustment. Subscales include Emotional Symptoms, Conduct Problems, Hyperactivity-Inattention, Peer Problems, and Prosocial Behavior. A Total Difficulties score is also provided. Four different versions are administered based on the child's age. Higher raw scores on all scales except for Prosocial Behavior indicate more difficulties; higher raw scores on Prosocial Behavior indicate greater prosocial behavior.
Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) | 6 months post-injury
  Adaptive functioning is measured using the Vineland Adaptive Behavior Scales, Third Edition (Vineland-3). Parents complete items designed to assess their child's ability to perform day-to-day activities in the domains of Communication, Daily Living, and Socialization. Composite scores are computed for each domain, as well as a general Adaptive Behavior Composite. Higher standard scores indicate higher adaptive functioning.
Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) | 12 months post-injury
  Adaptive functioning is measured using the Vineland Adaptive Behavior Scales, Third Edition (Vineland-3). Parents complete items designed to assess their child's ability to perform day-to-day activities in the domains of Communication, Daily Living, and Socialization. Composite scores are computed for each domain, as well as a general Adaptive Behavior Composite. Higher standard scores indicate higher adaptive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Amery Treble, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is currently no IPD sharing plan in place. If the investigators choose to share IPD in the future, they will create an IPD sharing plan in consultation with the University of Pittsburgh Office of Sponsored Programs.

REFERENCES:
- [Derived] Treble-Barna A, Patronick J, Uchani S, Marousis NC, Zigler CK, Fink EL, Kochanek PM, Conley YP, Yeates KO. Epigenetic Effects on Pediatric Traumatic Brain Injury Recovery (EETR): An Observational, Prospective, Longitudinal Concurrent Cohort Study Protocol. Front Neurol. 2020 Jun 12;11:460. doi: 10.3389/fneur.2020.00460. eCollection 2020. PMID 32595586